CLINICAL TRIAL: NCT04529122
Title: A Registry to Collect Characteristics and Outcomes From Patients With Solid Tumors Profiled With a Next-Generation Sequencing Test (WAYFIND-R)
Brief Title: A Worldwide Cancer Registry Enrolling Participants Profiled With a Next-Generation Sequencing Test
Status: Recruiting | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: MX39897
Record Dates: First submitted 2020-08-25; First posted 2020-08-27 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Solid Tumours

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
WAYFIND-R is a registry that aims to capture high-quality real-world data linking next-generation sequencing, treatments and outcomes from cancer patients diagnosed with a solid tumour. The WAYFIND-R has three main overarching objectives: 1. To provide a platform to support the design and conduct of clinical and epidemiological research; 2. To develop an evidence-generation platform to better understand health outcomes and cancer care processes; and 3. To characterize the treatments and clinical course of solid tumor cancers in patients who have undergone NGS testing.

ELIGIBILITY:
Inclusion Criteria:

* Participant is an adult (according to the age of majority as defined by local regulations)
* Participant is currently diagnosed with any type of solid tumour cancer, at any stage of the disease, at the enrollment date (informed consent date)
* Participant has undergone NGS testing, no longer than 3 months prior to the enrollment date, irrespective of the availability of test results
* Informed consent has been obtained from the participant or legally authorized representative, as per local regulations

Exclusion Criteria:

-Participant has a prior or current diagnosis of haematological malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and Female adult participants who are diagnosed with solid tumour cancers (at any anatomical location) and at any stage of the disease who have undergone an NGS test.
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2020-08-27 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | From date of registry entry until death, for up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (137):
- Argentina (2):
  - Instituto Alexander Fleming, Buenos Aires
  - CEMIC, Buenos Aires
- Lkh-Univ. Klinikum Graz, Graz, Austria
- Brazil (5):
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Instituto do Cancer do Estado de Sao Paulo - ICESP, São Paulo, São Paulo
  - Hospital Alemao Oswaldo Cruz, São Paulo, São Paulo
  - D'or Instituto de Pesquisa e Educação, Rio de Janeiro
  - Beneficencia Portuguesa de Sao Paulo, São Paulo
- Canada (2):
  - Alberta Health Services, Calgary, Alberta
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
- Chile (2):
  - Centro de Oncología de Precisión, Las Condes
  - Centro de Cancer Pontificie Universidad Catolica de Chile, Santiago
- Colombia (6):
  - Fundación CTIC - Centro de Tratamiento e Investigación sobre Cáncer Luis Carlos Sarmiento Angulo, Bogota, D.C.
  - Fundacion Cardioinfantil, Bogotá
  - Organizacion Sanitas Internacional, Bogotá
  - Fundacion Clinica Valle del Lili, Cali
  - Instituto Cancerología Medellin, Medellín
  - Clinica ASTORGA, Medellín
- International Medical Center, Cairo, Egypt
- Estonia (3):
  - East Tallinn Central Hospital, Tallinn
  - North Estonia Medical Centre Foundation, Tallinn
  - Tartu Uni Hospital, Tartu
- France (22):
  - Chu Amiens - Picardie, Amiens
  - Hopital Jean Minjoz, Besançon
  - Centre Hospitalier de Béthune-Beuvry, Béthune
  - Chu Brest - Hôpital Morvan, Brest
  - Centre Francois Baclesse, Caen
  - Centre Hospitalier de Chauny, Chauny
  - Centre Jean Perrin, Clermont-Ferrand
  - Groupe Hospitalier Public Du Sud De L'Oise GHPSO, Creil
  - Centre hospitalier universitaire Dijon-Bourgogne, Dijon
  - Hôpital Franco-Britannique- Fondation Cognacq-Jay, Levallois-Perret
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - APHM, Marseille
  - Hopital de La Timone - CHU de Marseille, Marseille
  - Institut Régional du Cancer de Montpellier, Montpellier
  - Institut Curie, Paris
  - CH de Cornouailles, Quimper
  - Centre Eugene Marquis, Rennes
  - CHU Saint Etienne - Hôpital Nord, Saint-Etienne
  - Hôpital Privé de la Loire, Ramsay Saint Etienne, Saint-Etienne
  - CHI de Toulon - Hôpital Sainte Musse, Toulon
  - Gustave Roussy, Villejuif
- Germany (10):
  - HELIOS Klinikum Bad Saarow, Bad Saarow
  - DRK Kliniken Berlin, Berlin
  - Universitätsklinikum Halle (Saale), Halle
  - Asklepios Klinik Altona, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - SLK-Kliniken Heilbronn GmbH;Klinik für Innere Medizin III, Heilbronn
  - Praxis für Hämatologie, Onkologie und Palliativmedizin, Mönchengladbach
  - Klinikum am Steinenberg / Ermstalklinik, Reutlingen
  - Katharinenhospital Stuttgart, Stuttgart
  - Marien-Hospital Wesel, Wesel
- Greece (5):
  - General Hospital "G.Papanikolaou", Asvestochóri
  - Henri Dunant Hospital, Athens
  - Alexandras General Hospital of Athens, Athens
  - Metropolitan Hospital Fourth Oncology Clinic, Faliro
  - Bioclinic Thessaloniki, Thessaloniki
- Hungary (2):
  - Bács-Kiskun Vármegyei Oktatókórház, Kecskemét
  - Pécsi Tudományegyetem, Pécs
- India (8):
  - Manipal Hospital, Bangalore, Karnataka
  - HealthCare Global Enterprises Limited, Banglore, Karnataka
  - Tata Memorial Hospital, Mumbai, Maharashtra
  - MOC Cancer Care & Research Centre (Unit of Cellcure Cancer Centre Pvt Ltd), Mumbai, Maharashtra
  - Bhaktivedanta Hospital and research institute, Thane, Maharashtra
  - Max Super Speciality Hospital, New Delhi, National Capital Territory of Delhi
  - Apollo Hospitals, Chennai, Tamil Nadu
  - Indo-American Cancer Hospital & Research Center, Hyderabad, Telangana
- Ireland (5):
  - Mid-Land Regional Hospital Tullamore, CO Offaly
  - Adelaide & Meath Hospital, Dublin, Incorporating the National Children's Hospital, Dublin
  - St Vincent'S Uni Hospital, Dublin
  - St James's Hospital, Dublin
  - Beacon Hospital, Dublin
- Israel (2):
  - Hadassah University Hospital - Ein Kerem, Jerusalem
  - Sourasky / Ichilov Hospital, Tel Aviv
- Lebanon (3):
  - American University of Beirut - Medical Center, Beirut
  - Hotel Dieu de France, Beirut
  - Hammoud Hospital, Saida
- Mexico (3):
  - ONCARE Viaducto Napoles, Mexico City, Mexico CITY (federal District)
  - Clínica Integral Internacional de Oncología S de RL de CV, Puebla City, Mexico CITY (federal District)
  - The American British Cowdray Hospital/ Hospital Abc, Mexico City
- Philippines (3):
  - Cebu Doctors' University Hospital, Cebu City
  - Metro Davao Medical and Research Center, Davao City
  - St Lukes Medical Center, Quezon City
- Narodowy Instytut Onkologii im. M. Sklodowskiej-Curie, Warsaw, Poland
- Portugal (3):
  - Hospital da Luz, Lisbon
  - Hospital CUF Porto, Porto
  - IPO do Porto, Porto
- National Guard King Abdulaziz Medical City, Riyadh, Saudi Arabia
- Serbia (5):
  - University Hospital Medical Center Bezanijska kosa, Belgrade
  - Oncomed-System, Belgrade
  - SIRIUS Medical, Belgrade
  - Special hospital for internal diseases Vesalius, Belgrade
  - Oncology Institute of Vojvodina, Kamenitz
- Narodny Onkologicky Ustav, Bratislava, Slovakia
- Slovenia (2):
  - University Clinic Golnik, Golnik
  - Institute of Oncology Ljubljana, Ljubljana
- South Africa (4):
  - IATROS International, Bloemfontein
  - Linksfield Oncology Inc., Johannesburg
  - Medical Oncology Centre of Rosebank, Johannesburg
  - Wilgers Oncology Centre, Pretoria
- Spain (5):
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Complejo Hospitalario de Jaen-Hospital Universitario Medico Quirurgico, Jaén
  - Hospital Clinico Universitario Virgen de la Victoria;Servicio de Oncologia, Málaga
  - Hospital Universitario Miguel Servet, Zaragoza
- Taiwan (3):
  - Chang Gung Medical Foundation - Kaohsiung, Kaohisung
  - Taipei Veterans General Hospital, Taipei
  - Chung Gung Memorial Hospital, Taoyuan
- Thailand (2):
  - Chulalongkorn Hospital, Bangkok
  - Faculty of Med. Siriraj Hosp., Bangkok
- Turkey (Türkiye) (8):
  - Medicana International Zincirlikuyu Hospital, Istanbul, Enter Text
  - Memorial Ankara Hastanesi, Ankara
  - Trakya University Medical Faculty, Edirne
  - Ba?c?lar Medipol Mega Üniversite Hastanesi, Istanbul
  - Medicana International Atasehir Hospital, Istanbul
  - Medicana International Izmir Hospital, Izmir
  - Ac?badem Maslak Hastanesi Büyükdere, Sar?yer/?stanbul
  - Ac?badem Adana Hospital, Oncology Department, Seyhan/Adana
- United Arab Emirates (2):
  - Tawam Hospital, Al Ain City
  - Mediclinic City Hospital, Dubai
- United Kingdom (12):
  - Blackpool Victoria Hospital, Blackpool
  - Bristol Haematology and Oncology centre, Bristol
  - Royal Sussex County Hospital, Eastbourne
  - Royal Devon & Exeter Hospital, Exeter
  - Gloucestershire Royal Hospital, Gloucester
  - Royal Surrey County Hospital, Guildford
  - St Georges University Hospitals NHS Foundation Trust, London
  - Freeman Hospital, New Castle Upon Tyne
  - Mount Vernon Hospital, Northwood
  - Musgrove Park Hospital, Somerset
  - Kings Mill Hospital, Sutton in Ashfield
  - Torbay Hospital, Torquay
- Vietnam (3):
  - Hanoi Oncology Hospital, Hanoi
  - K hospital, Hanoi
  - Ho Chi Minh City Oncology Hospital, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Dienstmann R, Hackshaw A, Blay JY, Le Tourneau C. Core variables for real-world clinicogenomic data collection in precision oncology. ESMO Real World Data Digit Oncol. 2025 Feb 27;7:100117. doi: 10.1016/j.esmorw.2025.100117. eCollection 2025 Mar. PMID 41647341
- See also: Related Info — https://www.wayfind-r.com/